CLINICAL TRIAL: NCT05878119
Title: Effects of MIB-626 (β-Nicotinamide Mononucleotide) With and Without A High-Intensity Multi-Dimensional Exercise Training Program on Physical Performance, Muscle Bioenergetics, and Neuropsychological Performance in Highly Fit Young Adults
Brief Title: Effects of MIB-626 With and Without A High-Intensity Multi-Dimensional Exercise Training Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metro International Biotech, LLC (Industry)
Responsible Party: Principal Investigator, Shalender Bhasin, Principal Investigator, Professor of Medicine, Harvard Medical School Director, Research Program in Men's Health: Aging and Metabolism Co-Director, BWH Center for Transgender Health Director, Boston Claude D. Pepper Older Americans Independence Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIB-626-206
Record Dates: First submitted 2023-03-01; First posted 2023-05-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Healthy; Physically Fit Adults; Regularly Exercising Adults; MIB-626

STUDY DESIGN:
Intervention Model Description: This will be two center, randomized, double-blind, placebo-controlled, parallel group trial to determine whether βNMN, after its daily oral administration, is associated with a greater reduction in the UACR compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind in that the study participants and the study staff involved in outcomes assessments will be unaware of the intervention assignment. The randomization schedule will be masked from all study personnel except those specifically designated below.
  The unblinded study biostatistician The staff of the Investigational Drug Pharmacy Services. The DSMB, if requested
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Investigational Product - MIB 626 plus usual physical activity (MIB-626- UPA) (Active Comparator): The MIB-626 will be a GMP-grade microcrystalline solid NMN mixed with inert excipients (including microcrystalline cellulose) and compressed into tablets at a dose strength of 500 mg per tablet, enabling administration of the 1,000 mg twice daily using two tablets taken twice daily.
  Interventions: Drug: Investigational Product - MIB 626; Other: Usual Physical Activity
- Placebo plus usual physical activity (PL-UPA) (Placebo Comparator): Matching placebo tablets will be provided by the study's Sponsor, Metro International Biotech, LLC.
  Interventions: Drug: Placebo; Other: Usual Physical Activity
- MIB-626 plus standardized, progressive, high intensity, multidimensional exercise (MIB-626-Ex) (Active Comparator): The MIB-626 will be a GMP-grade microcrystalline solid NMN mixed with inert excipients (including microcrystalline cellulose) and compressed into tablets at a dose strength of 500 mg per tablet, enabling administration of the 1,000 mg twice daily using two tablets taken twice daily.
  Interventions: Drug: Investigational Product - MIB 626; Other: Standardized, progressive, high intensity, multidimensional exercise
- Standardized, progressive, high intensity, multidimensional exercise plus placebo (PL-Ex) (Placebo Comparator): Matching placebo tablets will be provided by the study's Sponsor, Metro International Biotech, LLC.
  Interventions: Drug: Placebo; Other: Standardized, progressive, high intensity, multidimensional exercise

INTERVENTIONS:
Drug: Investigational Product - MIB 626 — The MIB-626 will be a GMP-grade microcrystalline solid NMN mixed with inert excipients (including microcrystalline cellulose) and compressed into tablets at a dose strength of 500 mg per tablet, enabling administration of the 1,000 mg twice daily using two tablets taken twice daily.
  Other Names: Investigational Product
  Arms: Investigational Product - MIB 626 plus usual physical activity (MIB-626- UPA); MIB-626 plus standardized, progressive, high intensity, multidimensional exercise (MIB-626-Ex)
Drug: Placebo — Placebo - Participants randomized to placebo will receive Matching placebo tablets will be provided by Metro International Biotech, LLC
  Arms: Placebo plus usual physical activity (PL-UPA); Standardized, progressive, high intensity, multidimensional exercise plus placebo (PL-Ex)
Other: Standardized, progressive, high intensity, multidimensional exercise — Participants will be asked to perform high intensity, standardized, progressive, multidimensional exercise.
  Arms: MIB-626 plus standardized, progressive, high intensity, multidimensional exercise (MIB-626-Ex); Standardized, progressive, high intensity, multidimensional exercise plus placebo (PL-Ex)
Other: Usual Physical Activity — Participants will be asked to perform usual physical activity per listed in the protocol
  Other Names: Usual Physical Acitivty
  Arms: Investigational Product - MIB 626 plus usual physical activity (MIB-626- UPA); Placebo plus usual physical activity (PL-UPA)

SUMMARY:
A single-center, randomized, placebo-controlled study in community dwelling, healthy, regularly exercising, highly physically fit men and women, 19 to 40 years. Eligible participants will be randomized to receive either 1000 mg NMN or placebo twice daily for 10 weeks.

DETAILED DESCRIPTION:
The study participants will be screened for potential participation and those meeting eligibility criteria on screening will be offered participation in the study. 120 subjects will be block randomized in a 1:1:1:1 ratio, stratified by sex (male, female) and baseline VO2 max. Participants will be randomly assigned to one of four groups using a 2 by 2 factorial design: Group 1 - MIB-626 (MIB-626 - UPA) plus usual physical activity; Group 2 - standardized, progressive, high intensity, multidimensional exercise plus placebo (PL-Ex); Group 3 - MIB-626 plus standardized, progressive, high intensity, multidimensional exercise (MIB-626-Ex); Group 4 - placebo plus usual physical activity (PL-UPA).

ELIGIBILITY:
Inclusion Criteria:

1. Highly physically fit and familiar with high intensity exercise training, as indicated

   1. Engages in vigorous exercise regularly (4 or more days each week) for 30 minutes or longer and which includes elements of resistance exercise training
   2. Physically fit ascertained using Daniels' equation https://runsmartproject.com/calculator/, 5K time: ≤ 23.0 min, and/ or 10K time: ≤ 48.0 min These criteria will maximize the likelihood of including individuals with VO2max of at least 40 mL/kg/min.
2. Has a body mass index (BMI) between 18.5 and 32 kg/m2, inclusive
3. Willingness to engage in 10-weeks of intensive exercise training designed to improve aerobic capacity and endurance, muscle strength, power, and fatigability, anaerobic capacity, and body composition, and to reduce fatigue
4. Willing to not engage in additional exercise training if randomized to the progressive exercise group and willing to not change usual physical activity if assigned to the usual physical activity group
5. Is free from clinically significant medical problems as determined by the Investigator
6. Is capable of providing written informed consent.
7. Is willing and able to provide authorization for the use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act (HIPAA).

In addition, female participants must:

1. Not be pregnant and not planning to become pregnant over the next 6 months

Exclusion Criteria:

1. Has AST or ALT > 2 times the upper limit of normal
2. Hematocrit < 36% or > 50% for men, or < 35% to > 48% for women
3. Has a diagnosis of diabetes or is using diabetes medications or has an A1C > 6.4%
4. Serum creatinine > 2.0 mg/dL or eGFR <60 mL/min
5. Prohibited medications and substances:

   a. Use of any performance enhancing substance (anabolic steroids, rhGH, DHEA, androstenedione, or any other performance enhancing drug
6. Current use of opiates, amphetamine, cannabinoids and cocaine

   1. Use of any other dietary supplement during the course of the trial. Subjects who are using a supplement containing nicotinamide or niacin or nicotinamide riboside may be included if they agree to stop the supplement at least 2 weeks prior to randomization and agree not to use such supplement/s during the entire duration of the study.
   2. Initiation of a new pharmaceutical product during the preceding 3 months
7. Known allergy to niacin or nicotinamide mononucleotide
8. In the judgment of the study physician, the participant is unlikely to comply with the study protocol for any reason or it may not be safe to administer the study.
9. Competing in organized athletics (e.g., collegiate sports) or training in preparation for competition
10. Contraindications to magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). These include: a) electrical implants such as cardiac pacemakers b) ferromagnetic implants such as aneurysm clips, surgical clips, artificial hearts valves with steel parts, shrapnel or steel implants c) ferromagnetic objects such as jewelry or metal clips in clothing d) pre-existing history of claustrophobic reactions. (Some participants who cannot undergo MRI/MRS but can undergo other study procedures might be considered on a case-by-case basis)

For women only:

1. Pregnant or planning to get pregnant over the next 6 months
2. Use of oral contraceptives is allowed provided the contraceptive regimen was initiated at least 3 months before randomization and the participant agrees not to change the regimen during the course of the study. 6.3 Excluded Medications and Treatments

1. The ingestion of the following is prohibited during 14 days prior to Day 0 and for the duration of the intervention period:

* Multivitamin preparations that contain niacin or one of its metabolites
* Products that contain niacin, nicotinic acid, nicotinamide in any form, other than natural foods
* Herbal supplements 2. Treatment with another investigational drug, investigational device, or approved therapy for investigational use within 3 month is prohibited.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic capacity from baseline to week 11, identified as VO2 max measured during a standardized increasing work rate treadmill protocol | 11 Weeks
  To determine the effects of MIB-626 (microcrystalline β-Nicotinamide Mononucleotide), administered at a dose of 1000-mg twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on aerobic capacity, assessed as VO2 max measured during a standardized increasing work rate treadmill protocol, in community living, healthy, regularly exercising, highly physically fit, men and women, 19 to 40 years, inclusive.

SECONDARY OUTCOMES:
Change in endurance time from baseline to week 11, measured during a constant work rate test | 11 weeks
  To determine the effects of MIB-626, administered at a dose of 1000-mg twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training, on endurance time during a constant work rate test.
Change from baseline to week 11 in anaerobic threshold during CPXT | 11 weeks
  To determine the effects of MIB-626 administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on anaerobic threshold by assessing peak anaerobic power, average anaerobic capacity, rate of power decay, and fatigue index using the Wingate anaerobic power test.
Change in upper body muscle performance, assessed as change from baseline to week 10 | 10 weeks
  To determine the effects of MIB-626, administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on upper body muscle performance using the instrumented chest press machines (Keiser).
Change in lower body muscle performance, assessed as change from baseline to week 10 | 10 weeks
  To determine the effects of MIB-626, administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on lower body muscle performance using the instrumented Keiser leg press machines.
Change over the 10 weeks in performance scores on sustained-attention, reaction-timed task | 10 weeks
  To determine the effects of MIB-626, administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus using a standardized Psychomotor Vigilance Task test.
Change over 10 weeks in working memory and working memory capacity | 10 weeks
  To determine the effects of MIB-626, administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on working memory and working memory capacity during a standardized continuous performance task assessed by using the n back test
Change over 10 weeks in selective attention, target identification and response | 10 weeks
  • To determine the effects of MIB-626, administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on selective attention, target identification and response (delay in reaction time between congruent and incongruent stimuli) using the STROOP test.
Change over 10 weeks in total sleep time | 10 weeks
  To determine the effects of MIB-626 administered twice daily for 10 weeks, with and without a standardized multidimensional program of progressive high intensity exercise training on total sleep time measured using an Actigraph device
Change from baseline in insulin sensitivity | 10 weeks
  To determine the effects of MIB-626 on insulin sensitivity by assessing fasting glucose, insulin and a derived index of insulin sensitivity by using (HOMA-IR)
Changes from baseline in blood lipid profile | 10 weeks.
  To evaluate the physiologic effects of MIB-626 on blood lipid profile by assessing the levels of plasma lipids, free fatty acids, leptin, myostatin, and adiponectin in the blood.
Change from baseline in sleep latency | 10 weeks
  and without a standardized multidimensional program of progressive high intensity exercise training on sleep latency measured using an Actigraph

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared